CLINICAL TRIAL: NCT02338453
Title: Examining the Effects of a Combined Attention Bias Modification Treatment (ABMT) and Cognitive-Behavioral Group Therapy (CBGT) for Social Anxiety Disorder
Brief Title: Attention Bias Modification Treatment (ABMT) and Cognitive-Behavioral Group Therapy (CBGT) in Social Anxiety Disorder
Acronym: ABMT+CBGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yair Bar-Haim (Other)
Collaborators: Geha Mental Health Center (Other)
Responsible Party: Sponsor-Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TauGeha-001-15
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety; Attention Modification; Dot-Probe; GCBT
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification Treatment (Active Comparator): Participants will receive an attention bias modification protocol designed to divert attention away from socially-threatening stimuli via repeated trials of a dot-probe task.
  Interventions: Behavioral: Active Attention Bias Modification Treatment
- placebo-control condition (Placebo Comparator): Participants will receive an placebo control protocol using the same task and stimuli but not designed to change attention patterns
  Interventions: Behavioral: Placebo Attention Bias Modification Treatment

INTERVENTIONS:
Behavioral: Active Attention Bias Modification Treatment — Attention bias is modified using a dot-probe task. Each trial begins with a fixation cross presented in the center of the screen for 500 ms. Next, participants are presented with two stimuli depicting two faces of the same individual for 500 ms, either of two neutral faces or with one neutral face and one disgust face (i.e., the socially-threatening stimulus). Then, one of two optional probes appears in the location former occupied by one of the faces. Participants are instructed to discriminate as fast as possible between the two variants of the probe, without compromising accuracy, by pressing on two corresponding keys. The probe remains on the screen until the participant responds, after which the next trial commences. This protocol is designed to divert attention away from socially-threatening stimuli as in 80% of trials the probe appears in the location formerly occupied by the neutral face. The remaining 20% of trials include two neutral faces, with no predictive value
  Other Names: Active ABMT
  Arms: Attention Bias Modification Treatment
Behavioral: Placebo Attention Bias Modification Treatment — the Placebo ABMT is similar to the active ABMT except that this protocol is not designed to divert attention away from or toward socially-threatening stimuli as in 40% of trials the probe appears in the location formerly occupied by the neutral face and in 40% it appears in the location formally occupied by the threatening face. The remaining 20% of trials include two neutral faces
  Other Names: Placebo ABMT
  Arms: placebo-control condition

SUMMARY:
This RCT examines the effectiveness of Attention Bias Modification Treatment (ABMT) as an augment to Cognitive-Behavioral Group Treatment (CBGT) for Social Anxiety Disorder (SAD) in adults. It is expected that ABMT vs. control training condition would achieve better therapeutic outcomes as indicated reduction in symptoms.

Participants from three groups (estimated 40 patients) will be offered to participate in the study

DETAILED DESCRIPTION:
Outpatients seeking treatment for Social Anxiety Disorder (SAD) at Geha anxiety-disorders clinic will be randomized into two groups (ABMT+CBGT; placebo control+CBGT). One group will undergo an Attention Bias Modification Treatment (ABMT) aimed at diverting attention away from socially-threatening stimuli. The second group will receive a placebo-control not designed to affect attention. Both groups will also undergo a standard Cognitive-Behavioral Group Treatment (CBGT) comprising 18 weekly sessions of 1.5-hr duration (along the lines of Heimberg, Juster, Hope & Mattia 1995 and Clark & Wells 1995). Symptoms and attention bias measures will be taken at three time points: Pre-treatment, Post-treatment,and at 3-month follow-up.

The study includes the following steps: a) initial assessment of participants' psychopathology and symptom levels; b) attention bias measurement; c) 8 sessions of ABMT/placebo control delivered as part of the CBGT sessions; d) two booster ABMT/Placebo treatments will be delivered at sessions 13 and 16 of the CBGT protocol. e) post-treatment assessment will include symptom and attention bias assessments. Finally, f) a three-month follow up assessment.

The goal of the study is to to test the effectiveness of ABMT as an add-on to established CBGT protocol for social anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form
* Men and women between the ages of 18 and 60.
* Meeting a current diagnosis of Social Anxiety Disorder (SP) according to the DSM-IV
* A minimum of a 1-year duration of SP
* SP as the primary diagnosis: In cases of co-morbidity, SP will be deemed as the most distressing and clinically significant condition among the co-morbid disorders
* Stable pharmacotherapy: Participants receiving a pharmacological treatment who are taking a stable medication for at least 3 months before the beginning of CBGT.

Exclusion Criteria:

* Psychotic episode in the past or the present time.
* Co-morbidity with any neurological disorder (i.e., epilepsy, brain injury).
* Another psychotherapeutic treatment during the study.
* Usage of neuroleptic medication.
* Change in medication status during the study.
* Substantial usage of drugs or alcohol in the present time.
* Poor judgment capacity (i.e., children under 18 and special populations).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline - the Liebowitz Social Anxiety Scale - Diagnostic Interview (LSAS; Liebowitz, 1987) scores | post treatment (18 weeks) and 3-month follow up
  The LSAS is a 24-item scale, each item corresponding to a situation selected on the basis of clinical experience. Each item is rated on a severity scale ranging from 0 to 3 with regard to the passing week, measuring separately two components of social anxiety, specifically, fear/anxiety and avoidance of social interaction and performance situations. Although the assessor may request and ask for further detail and adjust the rating based on clinical experience, this option is not often exercised, and inter-rater agreement is not considered to be a relevant concern (Safren et al., 1999). It has been shown to have strong psychometric properties, including high internal consistency, strong convergent and discriminative validity and high test-retest reliability (Fresco et al., 2001; Heimberg et al., 1999)

SECONDARY OUTCOMES:
Change from baseline - the Social Phobia Inventory (SPIN; Connor et al., 2000) scores | post treatment (18 weeks) and 3-month follow up
  This is a 17-item self-report measure of social anxiety evaluating fear, avoidance and physiological discomfort. Each item is rated on scale ranging from 0 to 4 with a possible total score of 68. The SPIN has been used in clinical and nonclinical samples and its psychometric properties have been found to be sound (Connor et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Haggai Hermesh, PhD, Study Chair — Geha Mental Health Center
Locations (2):
- Israel (2):
  - Geha Mental Health Center, Petah Tikva
  - Tel-Aviv University, Tel Aviv

REFERENCES:
- [Background] Shechner T, Rimon-Chakir A, Britton JC, Lotan D, Apter A, Bliese PD, Pine DS, Bar-Haim Y. Attention bias modification treatment augmenting effects on cognitive behavioral therapy in children with anxiety: randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2014 Jan;53(1):61-71. doi: 10.1016/j.jaac.2013.09.016. Epub 2013 Oct 10. PMID 24342386